CLINICAL TRIAL: NCT03872518
Title: A Prospective Case Series Analysis of Initial Users of the Urovac Device
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Dignity Medical Solutions (Unknown); California Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Josh Pevnick, Assistant Professor of Medicine and Associate Director, Division of Informatics, Cedars-Sinai Medical Center
Other Study IDs: Pro00049729
Record Dates: First submitted 2019-03-07; First posted 2019-03-13 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Incontinence, Urinary
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Urovac — The Urovac is simply a regular plastic handheld urinal attached by tubing to a pump that evacuates urine to a reservoir. The Urovac is simply a regular plastic handheld urinal attached by tubing to a pump that evacuates urine to a reservoir. There is also a removable cloth-covered platform to reduce spills.

SUMMARY:
To document usage of the Urovac device among 30 initial users of the device in an acute rehabilitation facility, with analysis of whether and how patients benefitted, challenges encountered, and how benefits and challenges varied by patient type.

DETAILED DESCRIPTION:
The Urovac device holds the promise of improving care for many of these patients in a manner that may also significantly decrease costs. The aim of the study is to determine if this device may increase quality of life for patients by reducing urine spills, reducing falls by avoiding urgent situations where patients try to ambulate to the bathroom to avoid wetting sheets, reducing skin breakdown by avoiding urine spills, reducing excoriation of the glans penis, and reducing urinary tract infections.

The Urovac is simply a regular plastic handheld urinal attached by tubing to a pump that evacuates urine to a reservoir. There is also a removable cloth-covered platform to reduce spills. Allowing for the evacuation of urine from the urinal significantly improves its functionality. The Urovac can be left in place without risk of overflow or other spillage, such that a patient with UI requires less assistance. Improving the handheld urinal in this manner should thus allow for reduced usage of diapers, catheterization, and institutionalization. For patients with UI requiring hospitalization or institutionalization for other reasons, the Urovac could potentially reduce the associated labor and complication costs. Despite the clear clinical promise of the Urovac, it has only been used by a small number of patients to date. This study will document usage of the Urovac among 30 of the initial users of the device to better understand the benefits and challenges.

ELIGIBILITY:
Inclusion Criteria:

* Male patients who identify as having difficulty with functional urinary incontinence, such that it may be difficult to get to the toilet in time to urinate
* Patients age 18 or older

Exclusion Criteria:

* Patients with leg wounds or dysfunction which could be worsened by Urovac device placement
* Patients under age 18

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Study participants may be biologically female or male, but must have male genitalia (a penis) to participate.
Study Population: Males with urinary incontinence, defined as a condition in which patients have difficulty getting to and using the toilet to evacuate urine.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with Urovac device: 5-point scale | 24 hours after patient is given instructions on how to use Urovac device.
  Patient satisfaction with the Urovac device after two-hour use of the device, as measured by the statement: "I would recommend it to someone in a similar situation." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."
Patient perception of urine spills after using Urovac | 24 hours after patient is given instructions on how to use Urovac device.
  Patient perception of urine spills after using Urovac after two-hour use of the device, as measured by the statement: "Urovac helped to avoid urine spills ." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."
Patient perception of dignity preservation after using Urovac | 24 hours after patient is given instructions on how to use Urovac device.
  Patient perception of dignity preservation after using Urovac after two-hour use of the device, as measured by the statement: "Urovac helped preserve dignity." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."
Patient perception of ulcer prevention | 24 hours after patient is given instructions on how to use Urovac device.
  Patient perception of ulcer prevention after using Urovac after use of the device, as measured by the statement: "Urovac helped avoid decubitus ulcers, or helped keep them dry." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."
Patient perception of reduced risk of falls | 24 hours after patient is given instructions on how to use Urovac device.
  Patient perception of reduced risk of falls after using Urovac after use of the device, as measured by the statement: "Urovac helped reduce risk of falls related to getting to a toilet." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."
Patient perception of caregiver time spent on helping patient use bathroom | 24 hours after patient is given instructions on how to use Urovac device.
  Patient perception of caregiver time spent on helping patient use bathroom after using Urovac after use of the device, as measured by the statement: "Urovac helped save patient/caregiver time." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."
Clinician perception of Urovac effectiveness in avoiding foley catheterization or condom catheter | 24 hours after patient is given instructions on how to use Urovac device.
  Clinician perception of Urovac effectiveness in avoiding foley catheterization or condom catheter, as measured by the statement: "Urovac helped patient to avoid foley catheterization or condom catheter." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."
Clinician perception of Urovac effectiveness of decreasing development or severity of decubitus ulcers. | 24 hours after patient is given instructions on how to use Urovac device.
  Clinician perception of Urovac effectiveness of decreasing development or severity of decubitus ulcers, as measured by the statement: "Urovac helped patient with decubitus ulcers." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."
Clinician perception of Urovac effectiveness of decreasing risk of falls when going to the toilet | 24 hours after patient is given instructions on how to use Urovac device.
  Clinician perception of Urovac effectiveness of risk of falls when going to the toilet, as measured by the statement: "Urovac helped reduce risk of falls related to getting to a toilet." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."
Clinician perception of Urovac effectiveness of decreasing risk of hospitalization or skilled nursing facility | 24 hours after patient is given instructions on how to use Urovac device.
  Clinician perception of Urovac effectiveness of decreasing risk of hospitalization or skilled nursing facility, as measured by the statement: "Urovac helped patient avoid hospitalization or skilled nursing facility admission." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."
Clinician satisfaction with Urovac device: 5-point scale | 24 hours after patient is given instructions on how to use Urovac device.
  Clinician satisfaction with Urovac device, as measured by the statement: "I would recommend it to a physician colleague." The 5-point scale goes from 1-5, with 1 being "strongly disagree," 2 being "somewhat disagree," 3 being "neither agree nor disagree," 4 being "somewhat agree," and 5 being "strongly agree."

SECONDARY OUTCOMES:
Development of urinary tract infection after using Urovac | 24 hours after patient is given instructions on how to use Urovac device.
  Development of urinary tract infection after using Urovac, dichotomous measure (yes/no) measured by checking electronic health record for evidence of urinary tract infection after use of the device.
Average hours of daily use of Urovac by patient | 24 hours after patient is given instructions on how to use Urovac device.
  Average hours of daily use of Urovac by patient

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Pevnick, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- California Rehabilitation Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grigoryan L, Abers MS, Kizilbash QF, Petersen NJ, Trautner BW. A comparison of the microbiologic profile of indwelling versus external urinary catheters. Am J Infect Control. 2014 Jun;42(6):682-4. doi: 10.1016/j.ajic.2014.02.028. PMID 24837121